CLINICAL TRIAL: NCT04922619
Title: Evaluation of the Impact of a Tonotopy Based Fitting on the Speech and Musical Perception in New Cochlear Implanted Subjects. Prospective Randomized Crossover Study.
Brief Title: Study of Music and Speech Perception in New Cochlear Implanted Subjects Using or Not a Tonotopy Based Fitting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MED-EL Elektromedizinische Geräte GesmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: MED_EL_tonofit_Rennes_study
Record Dates: First submitted 2021-06-02; First posted 2021-06-10 (Actual); Last update posted 2021-10-20 (Actual); Status verified 2021-10

CONDITIONS: Sensorineural Hearing Loss, Bilateral
Keywords: cochlear implant strategy; tonotopy based fitting
MeSH Terms: conditions — Hearing Loss, Sensorineural

STUDY DESIGN:
Intervention Model Description: Two arms A and B:
  Arm A: patient's fitting with default fitting --> 6 weeks use --> tests and patient's fitting with tonotopy based fitting --> 6 weeks use --> tests
  Arm B: patient's fitting with tonotopy based fitting --> 6 weeks use --> tests and patient's fitting with default fitting --> 6 weeks use --> tests
Who Masked: Participant, Investigator
Masking Description: Double blind study: the patient and the investigator don't know the fitting.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cochlear Implant (CI) with default fitting then tonotopy based fitting (Active Comparator): Cochlear Implant with default fitting first during 6 weeks then with tonotopy based fitting during 6 weeks
  Interventions: Device: tonotopy based fitting then default fitting; Device: default fitting then tonotopy based fitting
- Cochlear Implant (CI) with tonotopy based fitting then default fitting (Active Comparator): Cochlear Implant with tonotopy based fitting during 6 weeks then with default fitting during 6 weeks
  Interventions: Device: tonotopy based fitting then default fitting; Device: default fitting then tonotopy based fitting

INTERVENTIONS:
Device: tonotopy based fitting then default fitting — Cochlear implant with default fitting then tonotopy based fitting
Device: default fitting then tonotopy based fitting — Cochlear implant with tonotopy based fitting then default fitting

SUMMARY:
Main objective:

Show the superiority of tonotopy based fitting strategy compared to default fitting strategy on the perception speech in noise.

Secondary objectives:

Show the superiority of tonotopy based fitting strategy compared to default fitting strategy on the perception of musical elements (contour test).

Show the non inferiority of tonotopy based fitting strategy compared to default fitting strategy on the perception of speech elements in quiet.

Show the superiority of tonotopy based fitting strategy compared to default fitting strategy on the qualitative preference for the listening of musical pieces.

DETAILED DESCRIPTION:
Introduction: Cochlear implantation allows the rehabilitation of profound bilateral deafness, restoring speech perception and verbal communication when the traditional hearing aid no longer provides satisfactory hearing gain (Nimmons et al.).

A cochlear implant includes an electrode array and its functioning is based on the principle of cochlear tonotopy: each electrode encodes a frequency spectrum according to its position in the cochlea (high frequencies are assigned to the basal electrodes and low frequencies to the apical electrodes).

The cochlear implant thus breaks down the frequency spectrum into a number of frequency bands via bandpass filters corresponding to the number of electrodes in the implant. During the fitting these bands can be modified by the audiologist.

The fitting software developed by the manufacturers proposed a default fitting with a lower limit between 100 and 250 Hz according to the brands and an upper limit of about 8500 Hz. The frequency bands assigned to each electrode follow a logarithmic scale with the high frequencies for the basal electrodes and the low frequencies for the apical electrodes. This distribution takes into account the number of active electrodes but does not take into account the anatomy and the natural cochlear tonotopy specific to each patient.

Several studies have analyzed the anatomical variations of the cochlear dimensions: size of the cochlea and the ratio between the contact surfaces of the electrodes with the cochlea are variable from one patient to another (Stakhovskaya O et al., P. Pelliccia et al.).

The insertion depth during surgery is also variable due to parameters related to the patients as well as to the operator, which seems to impact the understanding of speech in noise (Deep electrode insertion and sound coding in cochlear implants - Ingeborg Hochmair et al.).

Mathematical algorithms have recently been developed to estimate the cochlear tonotopy of each patient from a CT scan assessment (Jiam et al., Sridhar et al.). CT imaging of the implanted ear combined with 3D reconstruction software, provides cochlear length measurements (Cochlear length determination using Cone Beam Computed Tomography in a clinical setting - Würfel et al .) Using this approach it is possible to measure the position of each electrode relative to the cochlear apex. These measurements are applied to the modified Greenwood equation to obtain the tonotopic frequency for each electrode and to determine for each patient a fitting based on the tonotopy of each electrode.

Main objective:

Show the superiority of tonotopy based fitting strategy compared to default fitting strategy on the perception speech in noise.

Secondary objectives:

Show the superiority of tonotopy based fitting strategy compared to default fitting strategy on the perception of musical elements (contour test).

Show the non inferiority of tonotopy based fitting strategy compared to default fitting strategy on the perception of speech elements in quiet.

Show the superiority of tonotopy based fitting strategy compared to default fitting strategy on the qualitative preference for the listening of musical pieces.

Plan of the study:

It is a prospective open monocentric randomized crossover study: measures will be done on the patient at 6 weeks and 12 weeks post-activation.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient (>= 18 years old) speaking French
* Patient who fulfils the criteria for cochlear implantation

Exclusion Criteria:

* retro-cochlear pathology: auditory neuropathy, vestibular schwannoma
* patient with residual hearing < 60 dB HL at 250 Hz and < 80 dB HL at 500 Hz

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2021-06-10 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
speech recognition in noise | at 6 weeks post-activation
  The speech recognition in noise is evaluated with syllabic list of 40 phonemes. The patient has to recognize 20 syllables. The phonemes are scored: each good answer is scored 1 yielding a total between 0 and 1 (or 0% and 100%). Signal-noise-ratios of 9, 6, 3 and 0 dB will be tested with speech at 65 dB SPL.
speech recognition in noise | at 12 weeks post-activation
  The speech recognition in noise is evaluated with syllabic list of 40 phonemes. The patient has to recognize 20 syllables. The phonemes are scored: each good answer is scored 1 yielding a total between 0 and 1 (or 0% and 100%). Signal-noise-ratios of 9, 6, 3 and 0 dB will be tested with speech at 65 dB SPL.

SECONDARY OUTCOMES:
speech recognition in quiet | at 6 weeks post-activation
  The speech recognition in quiet is evaluated with syllabic list of 40 phonemes. The patient has to recognize 20 syllables. The phonemes are scored: each good answer is scored 1 yielding a total between 0 and 1 (or 0% and 100%).
speech recognition in quiet | at 12 weeks post-activation
  The speech recognition in quiet is evaluated with syllabic list of 40 phonemes. The patient has to recognize 20 syllables. The phonemes are scored: each good answer is scored 1 yielding a total between 0 and 1 (or 0% and 100%).
Melodic contour test | at 6 weeks post-activation
  The test stimuli of the melodic contour test (Galvin et al. 2007) are melodic contours composed of 5 notes of equal duration whose frequencies correspond to musical intervals. Nine distinct musical patterns have to be identified by the patient. Each good answer is scored 1 yielding a total between 0 and 1 (or 0% and 100%).
Melodic contour test | at 12 weeks post-activation
  The test stimuli of the melodic contour test (Galvin et al. 2007) are melodic contours composed of 5 notes of equal duration whose frequencies correspond to musical intervals. Nine distinct musical patterns have to be identified by the patient. Each good answer is scored 1 yielding a total between 0 and 1 (or 0% and 100%).
Qualitative measure of music | at 6 weeks post-activation
  The Gabrielsson scale (1988) is used to evaluate perceived sound quality as a multidimensional phenomenon, that is composed of a number of separate perceptual dimensions. Eight perceptual dimensions are evaluated: clarity, fullness, brightness vs dullness, hardness/sharpness vs softness, spaciousness, nearness, extraneous sound, loudness.
  Visual analog scales (VAS) are used for each dimension and the patient has to score the dimension on a 10 cm VAS (between 0 to 10).
Qualitative measure of music | at 12 weeks post-activation
  The Gabrielsson scale (1988) is used to evaluate perceived sound quality as a multidimensional phenomenon, that is composed of a number of separate perceptual dimensions. Eight perceptual dimensions are evaluated: clarity, fullness, brightness vs dullness, hardness/sharpness vs softness, spaciousness, nearness, extraneous sound, loudness.
  Visual analog scales (VAS) are used for each dimension and the patient has to score the dimension on a 10 cm VAS (between 0 to 10).

CONTACTS AND LOCATIONS:
Overall Officials: Benoit Godey, Pr, Principal Investigator — Rennes University Hospital
Locations (1):
- CHU Rennes, Rennes, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Creff G, Bernard-Le Liboux N, Coudert P, Bourdon H, Pean V, Wallaert N, Lambert C, Godey B. Tonotopic and Default Frequency Fitting for Music Perception in Cochlear Implant Recipients: A Randomized Clinical Trial. JAMA Otolaryngol Head Neck Surg. 2024 Nov 1;150(11):960-968. doi: 10.1001/jamaoto.2024.2895. PMID 39264640